CLINICAL TRIAL: NCT05330663
Title: High Energy Low Protein Renal Formula as Meal Replacement in Predialysis CKD Patients
Brief Title: Low Protein Renal Formula as Meal Replacement in Predialysis CKD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Fresenius Kabi Taiwan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SF20045B
Record Dates: First submitted 2022-03-26; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Oral nutrition supplement
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Low protein diet with Fresubin® renal
  Interventions: Dietary Supplement: Low protein diet with Fresubin® renal
- Standard of care (Other): Low protein diet with normal food
  Interventions: Other: Low protein diet with normal food

INTERVENTIONS:
Dietary Supplement: Low protein diet with Fresubin® renal — Low protein diet with Fresubin® renal Dosage: 1 bottle per day as a replacement for one regular meal. All patients will get individualized dietary counseling aimed at achieving a protein intake of 0.6-0.8 g/kg actual body weight/day and an energy intake of 30-35 kcal/kg actual body weight.
  Arms: Intervention group
Other: Low protein diet with normal food — All patients will get individualized dietary counseling aimed at achieving a protein intake of 0.6-0.8 g/kg actual body weight/day and an energy intake of 30-35 kcal/kg actual body weight/day.
  Arms: Standard of care

SUMMARY:
A high energy and low protein renal formula tailored for the specific needs of pre-dialysis CKD patients.

DETAILED DESCRIPTION:
Previous studies indicated that low-protein formula nutritional supplements may improve compliance with an LPD and are beneficial in the management of pre-dialysis CKD patients

This study will evaluate the suitability of the disease-specific enteral formula Fresubin® renal in predialysis chronic kidney disease patients.

ELIGIBILITY:
Inclusion criteria:

* Chronic kidney disease stage 4-5 (eGFR <30 mL/min/1.73m2)
* Age: 20-80 years
* Patients on low protein diet (0.6-0.8 g protein/kg/d) for at least 3 months
* Written informed consent

Exclusion criteria:

* Dialysis or planned start of dialysis within next 3 months
* Patients awaiting kidney transplantation
* BMI <18 and >30 kg/m2
* Malnourished patients with albumin levels less than 3 g/dL who need additional supplementation of calories and nutrients
* Severe liver disease, malignant disease, infectious disease
* Existing gastrointestinal diseases or pathological findings, which do not allow EN, e.g. intestinal atony, ileus, acute upper GI bleeding, shock, or malabsorption, e.g. inflammatory bowel disease, pancreatic disease, or previous surgical GI resection
* Severely impaired gastrointestinal function, i.e. severe constipation or acute diarrhea (≥ 3 loose or watery stools per day)
* Dysphagia or high aspiration risk
* Relevant CNS and/or psychiatric disorders
* Known allergic reaction or intolerance to any of the ingredients of the study product
* Planned surgery or hospitalization during study period
* Suspicion of drug abuse
* Patients unable to follow study instructions or keeping a dietary diary
* Pregnant or lactating women
* Participation in another clinical trial with an investigational product within 30 days prior to start of study or during the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Change of body weight | baseline to week 4
  Body weight measured in kilograms

SECONDARY OUTCOMES:
Change 3-day dietary record | baseline to week 4
  Total energy intake,3 macronutrients (carbohydrates, protein and lipids) and micronutrients
Change body composition | baseline to week 4
  Body composition measured by bioelectrical impedance analyses
Change of renal fuction | baseline to week 4
  blood urea nitrogen,serum creatinine and estimated glomerular filtration rate
Change of electrolytes | baseline to week 4
  Sodium,potassium,calciam,phosphorus and magnesium in the blood
Safety and compliance. | baseline to week 4
  gastrointestinal symptoms measured by questionnaire
Change in lipid analysis | baseline to week 4
  Change of cholesterol ,triglyceride ,and LDL-cholesterol in the blood
Change of Body Mass Index (BMI) levels | baseline to week 4
  BMI was calculate by body weight (kg) divided by the square of the height (m^2)
Change of waist circumference levels | baseline to week 4
  Waist circumference was measured by a tape
Change of grip strength levels | baseline to week 4
  hand grip strength was measured by grip strength device
Change of CRP | baseline to week 4
  Change of CRP in the blood
Change of nutrition status in blood test | baseline to week 4
  Serum albumin, pre-albumin, total protein, uric acid
Change of daily protein intake | baseline to week 4
  24-hour urine estimated protein intake with Maroni formula

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsu Chen, MDPHD, Principal Investigator — Division of Nephrology in Taichung Veterans General Hospital
Locations (1):
- Taichung Verterans General Hospital Taichung, Taichung, ROC, Taiwan